CLINICAL TRIAL: NCT04521881
Title: Intramuscular Tranexamic Acid for the Treatment of Symptomatic Mild Traumatic Brain Injury in Older Adults: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Clinical Randomisation of an Anti-fibrinolytic in Symptomatic Mild Head Injury in Older Adults
Acronym: CRASH-4
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-KEP-456; 2020-003391-40 (EudraCT Number)
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury, tranexamic acid, older adults
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: A randomised, double blind, placebo controlled trial among 10,000 older adults with mild traumatic brain injury.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be done by an independent clinical trials supply company. It will involve the removal of the original manufacturer's label and replacement with the clinical trial label bearing the randomisation number, which will be used as the pack identification. Apart from the randomisation number, all pack label texts will be identical for tranexamic acid and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): A single dose of Tranexamic acid 500mg given by intramuscular injection
  Interventions: Drug: Tranexamic Acid 500 MG
- Placebo (Placebo Comparator): One Injection of the placebo which is 10 mL Sodium Chloride (0.9%)
  Interventions: Drug: Tranexamic Acid 500 MG

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — given once as an intramuscular injection

SUMMARY:
Tranexamic acid (TXA) reduces head injury deaths. The CRASH-4 trial aims to assess the effects of early intramuscular TXA on intracranial haemorrhage, disability, death, and dementia in older adults with symptomatic mild head injury

DETAILED DESCRIPTION:
TXA reduces bleeding by inhibiting the enzymatic breakdown of fibrin blood clots. Results from randomised trials (CRASH-3 and NCT01990768) show that early treatment with TXA (given intravenously) reduces head injury deaths (pooled RR 0.89, 95% CI 0.80-0.99). In the CRASH-3 trial, the reduction in head injury deaths with TXA was largest in patients with mild and moderate head injuries, particularly if patients were treated soon after injury. However, the CRASH-3 trial included mild TBI patients only if they had intracranial bleeding on CT scan. It is uncertain whether the results apply to mild TBI patients more generally. CRASH-4 is a randomised, double blind, placebo-controlled trial in symptomatic mild TBI in about 10,000 older adults. The pilot phase will include about 500 patients. The trial aims to provide reliable evidence about the effects of early intramuscular TXA on intracranial haemorrhage, disability, death, and dementia in older adults with symptomatic mild head injury.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older (actual or estimated)
* History or evidence of head injury (e.g. laceration, bruise, swelling or pain in head or face)
* GCS ≥ 13
* Has one or more of the following:

  1. has or had any impaired consciousness (loss of consciousness, amnesia, or confusion)
  2. nausea or vomiting
* Within 3 hours of injury (do not include if interval cannot be estimated e.g. patient unable to confirm time of fall or patient found on floor after an unwitnessed fall and home alone)
* Not living in a nursing home, mental health institution or prison
* Patient will be conveyed to or is admitted to a participating hospital

Exclusion Criteria:

- TXA not clearly indicated (e.g. major bleeding) or contraindicated (e.g. suspected stroke)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2021-04-18 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Emergency department discharge | within 24 hours
  discharge

SECONDARY OUTCOMES:
Intracranial bleeding on CT scan | within 48 hours
  any bleeding on the last scan conducted within 48 hours of randomisation
Head injury related death | within 48 hours
  In-hospital head injury-related death within 48 hours of injury
All cause mortality | within 28 days
  Cause of death will be described
Disability | within 28 days
  The Barthel scale will be used to assess functional disability
Global assessment of ability to self-care | within 28 days
  Scale of 1 to 5
Neurosurgery | within 28 days
  receipt of neurosurgery and type
Days in ICU | within 28 days
  Number of days
Re-admission to hospital | within 28 days
  readmission after discharge
Vascular occlusive events | within 28 days
  pulmonary embolism, myocardial infarction, deep vein thrombosis and stroke
Seizures | within 28 days
Intramuscular injection site reaction | within 28 days
  frequency and type of reactions
Pneumonia | within 28 days
Adverse events | within 28 days
  Any untoward medical occurrence (other than pre-specified outcomes)
Dementia | 1 year
  The occurrence of all-cause dementia will be determined 12 months after randomisation. Dementia will be identified through linkage to routinely collected health-care data.

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Shakur-Still, Study Chair — London School of Hygiene and Tropical Medicine; Ian Roberts, Study Chair — London School of Hygiene and Tropical Medicine
Locations (2):
- United Kingdom (2):
  - The Royal London Hospital, London
  - St George's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared publicly when all planned analyses are completed by the CRASH-4 Trial Collaborators. This will be hosted on freebird.lshtm.ac.uk
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Totally anonymised data (without random allocation, patient, country and site identifiers) will be freely available.Where random allocation codes, country/site identifiers are requested, appropriate pre-specified analysis plan will need to be submitted to the Trial Management Group for review and if necessary, appropriate Ethics Committee approval will be required.
URL: http://freebird.lshtm.ac.uk

REFERENCES:
- See also: Trial website — https://crash4.lshtm.ac.uk
- See also: TXA background information — http://txacentral.lshtm.ac.uk